CLINICAL TRIAL: NCT01327261
Title: Fasting Comparative Bioavailability of Two Tablet Formulations of Levodopa /Benserazide in Healthy Volunteers: A Single- Dose Randomized- Sequence, Open -Label Crossover Study
Brief Title: Fasting Comparative Bioavailability of Two Tablet Formulations of Levodopa /Benserazide in Healthy Volunteers
Acronym: PHOE10903
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Buenos Aires (Other)
Collaborators: Laboratorios Phoenix S.A.I.C.y F. (Unknown)
Responsible Party: Guillermo Di Girolamo, Buenos Aires University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Phoenix-Evoser (PHOE 1-0903)
Record Dates: First submitted 2011-03-28; First posted 2011-04-01 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2011-03

CONDITIONS: Healthy Volunteers
Keywords: levodopa; benserazide; bioequivalence; pharmacokinetics; A Single - Dose; Randomized- Sequence; Open -Label Crossover Study
MeSH Terms: interventions — benserazide, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levodopa + benserazide (test formulation) (Experimental): A randomized-sequence, open-label, 2-period crossover study assessing relative bioavailability of two drug products containing the association levodopa + benserazide.
  Interventions: Drug: Levodopa + benserazide
- Levodopa + benserazide (reference formulation) (Active Comparator)
  Interventions: Drug: Levodopa + benserazide

INTERVENTIONS:
Drug: Levodopa + benserazide — Single oral dose of either Experimental or Active Comparator. Levodopa 200 mg/benserazide 50 mg tablets,with 200 mL of water.

SUMMARY:
A group of 24 healthy volunteers receive one tablet of an association of levodopa 200 mg and benserazide 50 mg corresponding to two drug products: a test formulation (Evoser ®; Phoenix S.A.I.C. y F., Buenos Aires, Argentina) and a reference formulation (Madopar ®; Roche Pharma, Switzerland) to assess their relative bioavailability. After administration of each formulation 17 blood samples are taken and levodopa is measured by HPLC. Pharmacokinetic parameters (AUC, Tmax and Cmax) are compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian Argentinean males and females volunteers aged 21 to 50 years with a body mass index from 19 to 27 kg/m2 were enrolled in this study.
* All volunteers provided written informed consent prior to study initiation.

Exclusion Criteria:

* History of cardiovascular, hepatic, renal, psychiatric, neurologic, hematologic, or metabolic disease
* Drug or alcohol abuse within 2 years before the start of the study
* Smoking
* HIV, hepatitis B, or hepatitis C infection
* Consumption of any prescribed or over-the-counter drug within 2 weeks before the study or
* Participation in a similar study within the past 6 months. Female subjects were not to be pregnant, planning to become pregnant, or breastfeeding at the time of the study, and were required to use an effective method of contraception (intrauterine device or hormonal method) throughout the study.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Comparison of Area Under the Curve and Peak Concentration of plasma levodopa reached after two different drug products containing levodopa + benserazide | Blood samples are collected up to 6 hours after dosing. (day 1)
  In order to comply with Argentine regulation for marketing approval this study includes 24 healthy volunteers to investigate whether the relative bioavailability of the test formulation met the regulatory criterion for the assumption of bioequivalence to the branded formulation. After dosing with each formulation, 17 blood samples are taken to measure plasma levodopa concentration by HPLC. With plasma concentration values, pharmacokinetic parameters are calculated and bioequivalence assessed with WinNonLin software.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | Clinical evaluation are performed up to 6 hours after dosing. (day 1)
  Volunteers are asked about any discomfort or unusual manifestation they feel. Vital signs are recorded at each sampling time.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Di Girolamo, MD, PhD, Principal Investigator — Buenos Aires University

REFERENCES:
- [Derived] Keller GA, Czerniuk P, Bertuola R, Spatz JG, Assefi AR, Di Girolamo G. Comparative bioavailability of 2 tablet formulations of levodopa/benserazide in healthy, fasting volunteers: a single-dose, randomized-sequence, open-label crossover study. Clin Ther. 2011 Apr;33(4):500-10. doi: 10.1016/j.clinthera.2011.04.012. PMID 21635995